CLINICAL TRIAL: NCT05584969
Title: Peer Support Groups Improve Infant Growth and Complementary Feeding Practices Among Refugees in Post-emergency Settlements in the West- Nile Region in Uganda
Brief Title: Peer Groups to Improve Infant Feeding Practices and Child Growth in Post-emergency Settlements in Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oklahoma State University (Other)
Collaborators: Lutheran World Federation (Unknown); Makerere University (Other); Nestlé Foundation for the Study of Problems of Nutrition in the World (Unknown)
Responsible Party: Principal Investigator, Joel Komakech, Principal Investigator, Oklahoma State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HS-19-2
Record Dates: First submitted 2022-10-12; First posted 2022-10-18 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Infant Malnutrition
Keywords: Infant complementary feeding; Refugees; Post-emergency settlements; Infant growth; Uganda; Maternal social support
MeSH Terms: conditions — Infant Nutrition Disorders

STUDY DESIGN:
Intervention Model Description: The intervention in Moms-only arm was run concurrently with a similar intervention in the Moms and Dads treatment arm. At the same time, the Control arm did not receive any intervention. Data were collected from all study arms at the same time during the study in order to compare the effect of the intervention in the treatment arms against the control.
Who Masked: Participant, Outcomes Assessor
Masking Description: The settlements that were assigned to the different study arms were at least 6 kilometers apart to reduce the possibility of spillover effects of the intervention. The participants in each study arm were blinded from 1) which other settlements were involved in the activities they were engaging in and 2) what activities were and who was involved in those activities within the other study arms. Data collectors/enumerators were blinded from the study arm assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Moms-only treatment arm (Experimental): In this treatment arm, 10 Care Groups comprised of only mothers (10 - 20 participants per group) engaged in the peer-led intervention that consisted of infant feeding guidelines [16], cooking demonstrations, and backyard farming demonstrations conducted over 10 months. The peer-led trainings lasted 60 - 90 minutes and were conducted every two weeks and supervised by a selected VHT.
  Interventions: Behavioral: Peer-led integrated nutrition education intervention delivered through Care Groups
- Moms and Dads treatment arm (Experimental): This treatment arm received a similar peer-led intervention to the Moms-only treatment arm, however, this arm comprised both moms and dads (a couple)
  Interventions: Behavioral: Peer-led integrated nutrition education intervention delivered through Care Groups
- Control arm (No Intervention): This was the comparison arm of the study. No intervention was provided to the participants of this arm. However, all study arm participants accessed the standard of care which was the routine health services delivered through the government health centers.

INTERVENTIONS:
Behavioral: Peer-led integrated nutrition education intervention delivered through Care Groups — The intervention comprised a peer-led integrated nutrition education training using the Care Group model developed by the TOPS program [13]. In the treatment arms, topics trained in the peer support groups included 1) group dynamics and social support, 2) infant feeding 3) adequate basic hygiene, 4) child growth and development, and 5) fathers' involvement. The training modules were adopted and modified from the community health extension workers (CHEWs) handbook [14] and the UNICEF IYCF counseling cards for community workers [15, 16]. Over the study, the intervention participants also engaged in cooking demonstrations targeting infant complementary foods preparation and backyard kitchen gardening.
  Arms: Moms and Dads treatment arm; Moms-only treatment arm

SUMMARY:
The goal of this randomized trial was to examine whether a peer-to-peer integrated intervention using Care Groups combining nutrition education and social support will improve infant growth and complementary feeding practices among refugees in the West-Nile region in Uganda. The aims of the study were to 1) determine the relationship of the intervention using the Care Group model on complementary feeding of infants, and 2) investigate the effects of a peer-led integrated nutrition education intervention using the Care Group model on growth among infants of refugees in Uganda.

Pregnant mothers (390) in their 3rd trimester were enrolled in a peer-led nutrition education intervention using the Care Group model. One treatment arm had moms only in the Care Groups while the other treatment arm had both moms and dads in the groups. Each study arm had a total of 10 Care Groups with 10-20 participants each. The control arm equally had 10 groups, however, did not receive the intervention. Each of the treatment arms participated in a biweekly integrated nutrition training hypothesized to effect behavioral change in infant feeding practices. The biweekly training started in March 2022 and ended in December 2022 with data collection at four-time points during the study (baseline, midline-I, II, and endline). Infant complementary feeding was evaluated using the World Health Organization & UNICEF guidelines. Infant growth was assessed using length-for-age z-scores, weight-for-age z-scores and weight-for-length z-scores. The Medical Outcomes Study (MOS) Social Support Index was used as a proxy to measure maternal social support. Effects of Care Group intervention on infant complementary feeding and growth were tested by study arm compared to the control arm.

DETAILED DESCRIPTION:
Brief introduction:

Low-and middle-income countries (LMICs) are "home" to most of the world's refugees, the majority of whom are women and children. Refugee children are vulnerable to undernutrition and poor health, and humanitarian agencies have highlighted child undernutrition as a key area for intervention during refugee situations. Complementary feeding of infants in refugee settlements remains inadequate; however, there is limited evidence on how to address these nutritional challenges in refugee settlements. In 2020, I conducted a year-long community-based randomized control trial among post-emergency settlements in the West Nile region in Uganda to examine whether an integrated nutrition education intervention delivered through Care Groups would improve infant feeding practices and growth in the post-emergency settlements in Uganda. The findings in this study may be used to design nutrition-sensitive programs and also inform policies targeting complementary feeding practices within post-emergency settlements in Uganda.

Study area:

The Adjumani district had been randomly selected among six districts and one city hosting refugees in the West Nile region. Initially, three settlements in the Adjumani district were randomly selected and assigned to the three arms of the study. Ayilo-I settlement was assigned as a Moms-only treatment arm, Pagirinya settlement was the Moms & Dads treatment arm while Nyumanzi settlement was the Control arm. During the recruitment of the participants, some fathers in the settlement (Pagirinya) assigned to the Moms & Dads treatment could not commit to participating in a year-long study because they had to move away from the settlement for jobs back to Juba, the capital of Sudan or nearby towns with more employment opportunities. Because of the limited number of participants in the Moms & Dads arm, a second randomization was done excluding the already selected settlements. Ayilo II was then selected as the other settlement to identify respondents for the Moms & Dads treatment arm. These settlements were at least six kilometers apart to reduce the possibility of spillover effects of the intervention. The village health team (VHTs) and health center midwife assistants supported the identification of pregnant mothers to be included in the study.

Sample size:

Prompt introduction of solid and semi-solid foods to infants was used as the primary outcome to determine the sample size because of its reliability as an indicator of infant and young child feeding practices. A sample size of 317 mothers was desired for strong power, based on calculations using GPower 3.1 software, with a type I error of 0.05, a power of 0.90, and an effect size of 0.2 to detect differences in the proportions of infants introduced to complementary foods at 6-8 months among the 3 study arms. A 23 percent loss during follow-up was estimated; thus, 390 women (15-49 years of age) in their third trimester of pregnancy were willing to participate. These women were enrolled before baseline data collection. Husbands were eligible to participate with their wives in the Moms & Dads treatment arm. A total of 321 mother-infant dyads completed the study.

Purposive sampling was used to identify pregnant women in their 3rd-trimester to be included in the study. VHTs and a midwife assistant from each settlement were contacted to support the respondent identification process due to their community roles in promoting health among expectant mothers. Identified pregnant women were crossmatched with an integrated maternity register from the health facility. Verification of pregnancy term was done with the help of the midwife assistant, VHT, and researcher by validating records in the antenatal card or maternity records book. Each of the chosen settlements formed the household sampling frame for one arm of the study; that is, each settlement had either: 1) Moms-only, 2) Moms & Dads combined, or 3) Control arm. The participants in the study were followed up from recruitment in January 2020 to the end of the study in December 2020.

Study Intervention:

A peer-led integrated nutrition education training program using the Care Group model developed by the USAID TOPS program comprised the intervention. We hypothesized that participants in the Care Group intervention would have better peer support and would have improved infant complementary feeding and growth compared to the participants in the control arm. For the intervention arms, topics trained in the peer support groups included 1) group dynamics and social support, 2) optimal breastfeeding and complementary feeding practices, 3) adequate basic hygiene, 4) child growth and development, and 5) fathers' involvement. The training messages were adopted and modified from the community health extension workers (CHEWs) training handbook and the United Nations Children Emergency Fund (UNICEF) infant and young feeding counseling cards for community workers. Selected images were included in each module for illustration adopted from the UNICEF-IYCF counseling cards for community workers.

Intervention groups:

In this study, Moms-only and Moms & Dads arms comprised the treatment arms also referred to as the intervention arms. The Control arm was the third study arm but did not receive the intervention. Each study arm comprised 10 groups with 10 - 20 members per group. For the study arms, volunteer leaders were selected within each group by the members. These leaders were referred to as peer group leaders. For the intervention arms, the peer group leaders were trained for five days using the same training tool that was to be used during the Care Group meetings. The peer group leaders were trained by identified village health team (VHTs) together with a nutrition and health educator from the Adjumani district. Only one refresher training for the peer group leaders was done during the entire study period even though at least two refresher trainings had been planned. The failure to conduct additional refresher training was due to measures undertaken to observe COVID-19 safety operating procedures (SoPs). Nevertheless, monthly feedback meetings were held for the peer group leaders with the VHTs to harmonize group meeting plans and address any challenges. These monthly meetings were also attended by the researcher. Each of the peer group leaders facilitated integrated nutrition training modules on a biweekly basis to the 10 to 20 group members identified in a Care Group to effect behavioral change. The group members were also encouraged to visit each other's homes as part of peer follow-up, however, caution to COVID-19 SoPs was emphasized.

Standard of care/ Control arm:

In this study, the Control arm did not receive the intervention. The Control arm comprised a standard of care that was expected to involve VHTs doing their routine work in the community supporting households concerning nutrition and health information for better maternal and child health. The GoU recommends having at least two VHTs in a village, which is between 50 and 70 households. These VHTs report directly to the nearest government health facility. Additionally, the VHTs are expected to promote government health programs and urge community members to access health-related services from government facilities.

Data Collection:

The structured questionnaire used for this study was adapted from the Demographic and Health Surveys and UNHCR standardized expanded nutrition surveys (SENS) guidelines. These two questionnaires have been widely accepted for sociodemographic, health, and nutrition data collection and related information for nationally representative samples and humanitarian populations. Additional questions to assess maternal social support were adopted from the medical outcomes study (MOS) social support scale. The final questionnaire was translated into Arabic, Dinka, and Madi languages which are widely spoken by the South Sudanese in the refugee settlements in Uganda. The questionnaires were then uploaded onto electronic tablets (Lenovo Tab P11) using the Qualtrics software (Offline version). The collected data with the electronic tablets were uploaded to Qualtrics cloud storage at the end of each data collection day. Only the principal investigator and research collaborators had access to the data as part of maintaining respondent data safety.

Four enumerators with a minimum qualification of an associate degree in nutritional science, social sciences, or related fields were recruited and trained on the questionnaire. Each enumerator was proficient in English and Arabic and one of the local languages (Madi, Nuer, or Dinka). A total of 10 households with women pregnant in their 3rd trimester were used to pretest the questionnaire in the Boroli refugee settlement. The Boroli refugee settlement where the pretesting was done was not among the settlements that were selected for the year-long study. The researcher was able to make minor revisions and adjustments mostly regarding the flow of questions in the Qualtrics software. Data collectors/enumerators were blinded from the study arm assignment. The collection of data/information from a single respondent was completed within 1 hour and 30 minutes. The data collection time points for this study were baseline (January), Midline-I (June), Midline-II (October), and Endline (December). At each data collection period, the participants were provided with a 1 kg bar of washing soap, 200 mL of vitamin A fortified cooking oil, and half a kilo each of iodized salt and sugar, all worth about 7,600 Ugx (1.5 USD) as compensation for participation in the study.

Ethical Considerations:

This study was approved by the Institutional Review Boards of the Uganda National Council of Science and Technology (SS 5038), Makerere University School of Health Science Research and Ethics Committee (SHSREC REF:2019-020), and Oklahoma State University (HS-19-2). Additional permission was acquired from the Office of the Prime Minister (OPM) Uganda (OPM/R/107). Informed consent was obtained from all respondents at recruitment for participation in the study, and before data collection during the study.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women of reproductive age (15 - 49 years) in their third trimester were eligible to participate in the study.
* Husbands were eligible to participate with their wives in the Moms & Dads treatment arm

Exclusion Criteria:

* Mothers whose antenatal records showed pregnancy complications were excluded from the study.
* Mothers who gave birth to premature infants, infants with congenital abnormalities, or whose infants died had the option of remaining in the study but were excluded from the final analyses.

Ages: 15 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 390 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2020-12-21 (Actual)

PRIMARY OUTCOMES:
Introduction of solid and semi-solid or soft foods (ISSSF) | through study completion, an average of 1 year
  Proportion of infants introduced to solid, semi-solid or soft foods at 6 months, continually breastfed and were between 6 - 8 months of age
Infant minimum dietary diversity scores (MDD) | through study completion, an average of 1 year
  Proportion of infants in the age category 6 - 23 months who consumed at least five food groups of the recommended eight in the past 24 hours. The food groups include - currently breastfed; roots and tubers; grains; flesh foods (meat, fish, poultry, and organ meats); legumes and nuts; dairy products; vitamin A-rich fruits and vegetables; eggs; other fruits and vegetables
Infant minimum meal frequency (MMF) | through study completion, an average of 1 year
  Proportion of infants in the age category 6 - 23 months who consumed solid, semi-solid or soft foods including snacks the recommended minimum number of times for both breastfed and non-breastfed infants. That is, a minimum of
  * 2 feedings for breastfed infants 6 - 8 months of age
  * 3 feedings for breastfed infants in the 9 - 23 months of age category
  * 4 feeding for non-breastfed infants in 6 - 23 months age category.
Infant minimum acceptable diet (MAD) | through study completion, an average of 1 year
  Proportions of infants who met composite indicator of optimal age specific frequency of meals and the adequate variety i.e.
  * Breastfed infants in the 6 - 23 months age range with adequate minimum dietary diversity and meal frequency in the past 24 hours
  * Non-breastfed infants within 6 - 23 months with adequate minimum dietary diversity and meal frequency in the past 24 hours in addition to at least two milk feeds
Eggs and or flesh foods consumption (EFF) | through study completion, an average of 1 year
  Proportion of infants between 6 - 23 months who consumed an egg or flesh foods in the previous day.
infant stunting | through study completion, an average of 1 year
  Length-for-age z-scores (LAZ)(The z-scores were calculated after subtracting the measured length of a child from the median value of the reference population and adjusted for sex and age). A cutoff of - 2 z-score indicates stunting.
infant underweight | through study completion, an average of 1 year
  Weight-for-age z-scores (WAZ)(The z-scores were calculated after subtracting the measured weight of a child from the median value of the reference population and adjusted for sex and age). A cutoff of - 2 z-score indicates underweight.
infant wasting | through study completion, an average of 1 year
  Weight-for-length z-scores (WAZ)(The z-scores were calculated after subtracting the measured length and weight of a child from the median value of the reference population and adjusted for sex and age). A cutoff of - 2 z-score indicates wasting.

SECONDARY OUTCOMES:
Maternal social support | through study completion, an average of 1 year
  Maternal social support was assessed with the medical outcomes study (MOS) social support scale [8]. A set of 19 questions with a five-point Likert scale was adapted from the MOS scale which has often been used in assessing social support. In this study, participants expressed the level of perceived support with responses ranging from "none of the time" (score of '1') to "all of the time" (score of '5'). The mother's perceived social support based on their total mean score was categorized into optimal (>4 and ≤5); moderate (>3 and ≤4), low (>2 and ≤3), and none or very low support (≤2)

CONTACTS AND LOCATIONS:
Overall Officials: Joel J Komakech, Ph.D., Principal Investigator — Oklahoma State University
Locations (1):
- Adjumani refugee settlements, Adjumani, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Any identifiers in the participants' data were removed in order to maintain the confidentiality of the participants. Other researchers will be able to access the cleaned dataset (csv or stata file type)with an excel file describing each of the variables. The researchers will also be able to access the study protocol to understand how the intervention was planned and implemented and the data collection process.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available from December 2021 to December 2031 (10 years)
Access Criteria: The study data will be shared on request from the principal investigator.

REFERENCES:
- [Background] UNHCR. Figures at a Glance: UNHCR, Geneva, Switzerland; 2020 [Available from: https://www.unhcr.org/en-us/figures-at-a-glance.html. Accessed January, 2022.
- [Background] Corbett M, Oman A. Acute Malnutrition in Protracted Refugee Situations: A Global Strategy. Geneva, Switzerland: UNHCR/WFP; 2006.
- [Background] Buscher D. New approaches to urban refugee livelihoods. Refuge: Canada's Journal on Refugees. 2013;28(2).
- [Background] Ministry of Health Uganda, Uganda Bureau of Statistics, Office of the Prime Minister Uganda, UNHCR. Food Security and Nutrition Assessment in Refugee Settlements and Kampala. Kampala: MOH and UNHCR Representation Office in Uganda; 2020.
- [Background] Style S, Tondeur M, Wilkinson C, Oman A, Spiegel P, Kassim IA, Grijalva-Eternod C, Dolan C, Seal A. Operational guidance on the use of special nutritional products in refugee populations. Food Nutr Bull. 2013 Dec;34(4):420-8. doi: 10.1177/156482651303400407. PMID 24605692
- [Background] Blanchet K, Ramesh A, Frison S, Warren E, Hossain M, Smith J, Knight A, Post N, Lewis C, Woodward A, Dahab M, Ruby A, Sistenich V, Pantuliano S, Roberts B. Evidence on public health interventions in humanitarian crises. Lancet. 2017 Nov 18;390(10109):2287-2296. doi: 10.1016/S0140-6736(16)30768-1. Epub 2017 Jun 8. PMID 28602563
- [Background] Marmot M, Friel S, Bell R, Houweling TA, Taylor S; Commission on Social Determinants of Health. Closing the gap in a generation: health equity through action on the social determinants of health. Lancet. 2008 Nov 8;372(9650):1661-9. doi: 10.1016/S0140-6736(08)61690-6. PMID 18994664
- [Background] Prudhon C, Benelli P, Maclaine A, Harrigan P, Frize J. Informing infant and young child feeding programming in humanitarian emergencies: An evidence map of reviews including low and middle income countries. Matern Child Nutr. 2018 Jan;14(1):e12457. doi: 10.1111/mcn.12457. Epub 2017 Jul 3. PMID 28670790
- [Background] WFP, UNHCR. Food Security and Nutrition Assessment in Refugee Settlements, Uganda 2017. Final Report. UNHCR SENS-Version 2. 2017.
- [Background] UNHCR. Uganda Comprehensive Refugee Response Portal 2020 [Available from: https://ugandarefugees.org/en/country/uga. Accessed February 2019
- [Background] Arikpo D, Edet ES, Chibuzor MT, Odey F, Caldwell DM. Educational interventions for improving primary caregiver complementary feeding practices for children aged 24 months and under. Cochrane Database Syst Rev. 2018 May 18;5(5):CD011768. doi: 10.1002/14651858.CD011768.pub2. PMID 29775501
- [Background] Waswa LM, Jordan I, Herrmann J, Krawinkel MB, Keding GB. Community-based educational intervention improved the diversity of complementary diets in western Kenya: results from a randomized controlled trial. Public Health Nutr. 2015 Dec;18(18):3406-19. doi: 10.1017/S1368980015000920. Epub 2015 Apr 10. PMID 25857703
- [Background] Food Security & Nutrition Network Social & Behavioral Change Task Force. Care Groups: A Training Manual for Program Design and Implementation. Washington D.C,: Technical and Operational Performance Support Program; 2014.
- [Background] Government of Uganda. Village Health Team: Participant Manual for Village Health Team Members. In: Ministry of Health, editor. Kampala, Uganda: Ministry of Health, Uganda; 2002.
- [Background] UNICEF. The Community IYCF Counselling Cards for Community Workers. In: United Nations Children's Fund, editor. Online. New York: UNICEF; 2020.
- [Background] UNICEF. The Community Infant and Young Child Feeding Counselling Package New York: UNICEF; 2022 [Available from: https://www.unicef.org/documents/community-iycf-package. Accessed March 2019.
- [Background] Turinawe EB, Rwemisisi JT, Musinguzi LK, de Groot M, Muhangi D, de Vries DH, Mafigiri DK, Pool R. Selection and performance of village health teams (VHTs) in Uganda: lessons from the natural helper model of health promotion. Hum Resour Health. 2015 Sep 7;13:73. doi: 10.1186/s12960-015-0074-7. PMID 26346431
- [Background] Macro International. Demographic and Health Surveys (DHS). https://dhsprogram.com/ 2018: Accessed November 2018.
- [Background] UNHCR. Standardised Expanded Nutrition Survey Guidelines for Refugee Populations (Version 3). 2019.
- [Background] Sherbourne CD, Stewart AL. The MOS social support survey. Soc Sci Med. 1991;32(6):705-14. doi: 10.1016/0277-9536(91)90150-b. PMID 2035047
- [Derived] Komakech JJ, Emerson SR, Cole KL, Walters CN, Rakotomanana H, Kabahenda MK, Hildebrand DA, Stoecker BJ. Care groups in an integrated nutrition education intervention improved infant growth among South Sudanese refugees in Uganda's West Nile post-emergency settlements: A cluster randomized trial. PLoS One. 2024 Mar 15;19(3):e0300334. doi: 10.1371/journal.pone.0300334. eCollection 2024. PMID 38489346
- [Derived] Komakech JJ, Emerson SR, Cole KL, Walters CN, Rakotomanana H, Kabahenda MK, Hildebrand DA, Stoecker BJ. A Peer-Led Integrated Nutrition Education Intervention through Care Groups Improved Complementary Feeding of Infants in Postemergency Settlements in the West-Nile Region in Uganda: A Cluster Randomized Trial. Curr Dev Nutr. 2023 Feb 3;7(3):100042. doi: 10.1016/j.cdnut.2023.100042. eCollection 2023 Mar. PMID 37181933